CLINICAL TRIAL: NCT00404859
Title: Monitoring Chronic Airway Inflammation in Children With Asthma and Cystic Fibrosis
Brief Title: FLAME: Airway Inflammation Monitoring in Asthma and Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: AstraZeneca (Industry); Cystic Fibrosis Foundation (Other)
Other Study IDs: MEC 05-114
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2005-12

CONDITIONS: Asthma; Cystic Fibrosis
Keywords: inflammometry; exhaled breath condensate; fractional exhaled nitric oxide; asthma; cystic fibrosis; monitoring; exacerbations; paediatric
MeSH Terms: conditions — Asthma; Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background By means of measurements of series of non-invasive inflammatory markers in exhaled breath (condensate), a reflection of inflammatory processes and oxidative stress, can be obtained. Thereby, these techniques could be important in monitoring asthma and CF lung disease in children. Fractional exhaled nitric oxide (FeNO) and inflammatory markers in exhaled breath condensate (EBC) reflect ongoing inflammation and oxidative stress in the airways. These markers have a promising capacity for monitoring diagnoses of CF and asthma lung disease.

Aim To study the course of inflammatory markers in time in children with asthma and CF, in stable periods and during pulmonary exacerbations. In addition, we study the ability of inflammatory markers to predict safe tapering of medical treatment in both populations.

1. To study the course of inflammatory markers in EBC during an exacerbation.
2. To study which IM are already elevated before a clinical exacerbation is evident and can predict exacerbations in time.
3. To study which inflammatory markers can predict safe discontinuation of antibiotics in children with CF, or tapering of inhaled corticosteroids in children with asthma.
4. To study the relationship between inflammatory markers in EBC, the severity and control of CF and asthma, the symptoms and lung function within patients will be analysed.

Methods Children with CF (n=30) and children with asthma (n=40) were recruited included from our outpatient clinic. During this longitudinal study patients visit the outpatient clinic were followed-up for 12 months; every two months during one year. patients visited our outpatient clinic. In addition to these standard visits, During exacerbations patients four extra visits were planned during an exacerbation. were asked to visit the University Hospital Maastricht four times. These additional visits were planned with a maximum of two times during the study. By means of a home monitor, children were asked to assess measurements of Besides measurements in the University Hospital, children measured forced expiratory volume in one second (FEV1) at home using a home monitor, to record medication use, and, to record presence and severity of pulmonary symptoms. Outcome parameters were: 1) FeNO assessment in exhaled air, 2) inflammatory markers in EBC, 3) lung function parameters, 4) specific questionnaires to assess asthma and CF control and severity, 5) data originating from the home monitor.

ELIGIBILITY:
Inclusion Criteria:

* Asthma is defined as a chronic inflammatory disorder, leading to recurrent episodes of wheezing, breathlessness, chest tightness, and/or coughing, based on variable airway obstruction [18]. Children with docter-diagnosed asthma known at the department of Paediatric Pulmonology, were recruited from the University Hospital Maastricht. Atopic and not atopic asthmatic children were allowed; treatment with inhalation corticosteroïd (ICS) was not obliged.
* Children known with CF were recruited from University Hospital Maastricht. CF was defined as a combination of typical clinical features and an abnormal sweat test (Chloride > 60 mM). CF lung disease was treated according to the CBO consensus ref. Main aspects of treatment were:

  * antibiotic treatment,
  * agents to promote airway secretion clearance, such as DNase,
  * bronchodilators, and,
  * physiotherapy. All alternations of medical therapy were allowed and accurately documented.

Exclusion Criteria:

* Diseases that may interfere with the results of the study (e.g. upper airway infection, cor vitium, anatomic abnormalities of the airway and other chronic inflammatory diseases, such as Morbus Crohn and rheumatoid arthritis),
* Mental retardation,
* Inability to perform measurements properly,
* Active smoking and,
* Use of the following medication: papaverin, sodium nitroprusside, angiotensin-converting enzyme (ACE) inhibitors, oxymetazoline, L-arginine, or nitric oxide synthase (NOS) inhibitors

Ages: 5 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70
Dates: Start 2006-01; Study Completion 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte M Robroeks, MD, Principal Investigator — Maastricht University Medical Center; Edward Dompeling, MD, PhD, Study Director — Maastricht University Medical Center; Quirijn Jöbsis, MD, PhD, Study Director — Maastricht University Medical Center
Locations (4):
- Netherlands (4):
  - Catharina Hospital, Eindhoven
  - University Hospital Maastricht, Maastricht
  - St Radboud Childrens Hospital, Nijmegen
  - Máxima Medical Centre, Veldhoven

REFERENCES:
- [Derived] Robroeks CM, van Berkel JJ, Jobsis Q, van Schooten FJ, Dallinga JW, Wouters EF, Dompeling E. Exhaled volatile organic compounds predict exacerbations of childhood asthma in a 1-year prospective study. Eur Respir J. 2013 Jul;42(1):98-106. doi: 10.1183/09031936.00010712. Epub 2013 May 3. PMID 23645402